CLINICAL TRIAL: NCT01631656
Title: Combination Finacea Gel and Vascular Nd:Yag Laser Therapy for Mild to Moderate Rosacea
Brief Title: Combination Gel and Vascular ND in Mild to Moderate Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00012702
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Rosacea
Keywords: Rosacea, Laser, Finacea Gel, Azelaic Acid,
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Azelaic Acid plus Laser (Experimental): Azelaic acid 15% twice daily on half the face for 6 weeks, plus laser treatment with Nd:Yag laser once at 2 weeks.
  Interventions: Drug: Azelaic acid; Device: Nd:Yag laser
- Laser only (Active Comparator): laser treatment on all face once at 2 weeks with no azelaic acid on one side of the face
  Interventions: Device: Nd:Yag laser

INTERVENTIONS:
Drug: Azelaic acid — 15% gel on half the face, twice daily, 6 weeks
  Other Names: Finacea gel
  Arms: Azelaic Acid plus Laser
Device: Nd:Yag laser — Treatment with Nd:Yag laser , once at Week 2.

SUMMARY:
This is a single center, open-label, split-face, prospective study of ten to fifteen subjects seeking vascular laser therapy for the treatment of mild to moderate rosacea. Subjects will be screened for eligibility for vascular laser therapy outside of the confines of this protocol. Once approved for laser, subjects will be screened for study enrollment and topical treatment of their rosacea at the Screening/Baseline visit. All subjects will receive Finacea 15% gel and will be instructed to apply the study drug to one half of the face, twice daily. Drug application will be modified just prior to and after the subjects' laser treatment to reduce irritation. Subjects will undergo Vascular Nd:Yag laser therapy to involved areas over the whole face two weeks after initiating Finacea treatment. Subjects will continue to use Finacea gel to one half of the face for the duration of the study.

DETAILED DESCRIPTION:
This is a single center, open-label, split-face, prospective study of ten to fifteen subjects seeking vascular laser therapy for the treatment of mild to moderate rosacea. Subjects will be screened for eligibility for vascular laser therapy outside of the confines of this protocol. Once approved for laser, subjects will be screened for study enrollment and topical treatment of their rosacea at the Screening/Baseline visit. All subjects will receive Finacea 15% gel and will be instructed to apply the study drug to one half of the face, twice daily. Drug application will be modified just prior to and after the subjects' laser treatment to reduce irritation. Subjects will undergo Vascular Nd:Yag laser therapy to involved areas over the whole face two weeks after initiating Finacea treatment. Subjects will continue to use Finacea gel to one half of the face for the duration of the study. Assessment of acneiform lesions, redness, and telangiectasias will be performed at Screening/Baseline, Week 2 (prior to laser treatment), and week 6/End of Study. Photography will be performed at Screening/Baseline and End of Study visits. Adverse events will be assessed at each visit, and a patient survey will be completed at Baseline and at Week 6/End of Study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with mild to moderate rosacea, age 18 and over, who agrees to participate and provide written consent.
* Have an Investigator Global Assessment of mild to moderate rosacea (IGA rating between 2 and 5 in the Investigator Global Assessment (Appendix B) and at least a "Mild" rating on the Telangiectasia Rating Scale
* Subjects must be eligible to undergo vascular laser therapy and have been previously approved for therapy.

Exclusion Criteria:

* Initiation or change in dose within 4 weeks of baseline of systemic anti-inflammatory medication which may influence study outcome.
* Use of topical therapy for rosacea within 2 weeks of baseline.
* Use of systemic corticosteroids within 4 weeks of baseline.
* Use of systemic retinoids within 6 months of baseline
* Presence of a concurrent medical condition or skin condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Amount of disease involvement that would require >60 gm of cream in a 6 week period.
* Subjects with known allergy or sensitivity to azelaic acid (Finacea®) gel or components therein, such as propylene glycol.
* Contraindication to vascular laser therapy, such as infections.
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Reliable methods of birth control are: abstinence (not having sex), oral contraceptives, intrauterine device (IUD), DepoProvera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dept of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azelaic Acid Left Side Plus Laser: Azelaic acid 15% twice daily for 6 weeks to the left side of the face, plus laser treatment with Nd:Yag laser once at 2 weeks.
  Azelaic acid: 15% gel, twice daily, 6 weeks
  Nd:Yag laser: Treatment with Nd:Yag laser to all the face, once at Week 2.
- Azelaic Acid Right Side Plus Laser: Azelaic acid 15% twice daily for 6 weeks to the right side of the face, plus laser treatment with Nd:Yag laser once at 2 weeks.
  Azelaic acid: 15% gel, twice daily, 6 weeks
  Nd:Yag laser: Treatment with Nd:Yag laser to all the face, once at Week 2.
Period: Overall Study
Arm/Group | Azelaic Acid Left Side Plus Laser | Azelaic Acid Right Side Plus Laser
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Left Side Plus Laser | Azelaic Acid Right Side Plus Laser | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: IGA of Improvement
Description: Investigator's Global Assessment of severity integrates all lesions for overall score. This measure is commonly used as a quick and simple way to quantify disease severity both for clinical studies and in a non-study clinic setting. Score ranges from 0 = Clear or "No inflammatory signs of rosacea" to 6 = "Severe inflammatory signs of rosacea."
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Azelaic Acid Plus Laser: Azelaic acid 15% twice daily for 6 weeks, plus laser treatment with Nd:Yag laser once at 2 weeks.
  Azelaic acid: 15% gel, twice daily, 6 weeks
  Nd:Yag laser: Treatment with Nd:Yag laser of half the face, once at Week 2.
- LASER ONLY: Laser treatment with no azelaic acid on one side of face
Arm/Group | Azelaic Acid Plus Laser | LASER ONLY
Number analyzed (Participants) | 10 | 10
units on a scale | 3.1 (1.2) | 3.5 (1.4)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Azelaic Acid Plus Laser: Azelaic acid 15% twice daily for 6 weeks on one side of the face, plus laser treatment with Nd:Yag laser once at 2 weeks.
Arm/Group | Azelaic Acid Plus Laser | Laser Only
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Plus Laser (N=10) | Laser Only (N=10)
herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes